CLINICAL TRIAL: NCT05900661
Title: The Effect of Myo-inositol, Somatropin, and DHEA on Poor Ovarian Responders Undergoing ICSI : an Open Label Randomized Clinical Trial.
Brief Title: The Effect of Myo-inositol, Somatropin, and DHEA on Poor Ovarian Responders
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: poor ovarian responders
Record Dates: First submitted 2023-06-04; First posted 2023-06-12 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Poor Responders
Keywords: Cetrorelix; DHEA; somatotropin; myo inositol
MeSH Terms: interventions — Inositol; Human Growth Hormone; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- myo-inositol (Experimental): will recive Inofolic (myo-inositol 600µgm + folic acid 0.2 mg) 2 capsules at the morning and 2 capsules at the evening on empty stomach for 12 weeks
  Interventions: Drug: myo-inositol
- Somatropin (Experimental): Somatropin (4 IU for 1month), SEDICO ,6th of october .Egypt. 1 s.c injection every 3 days for at least 1 month.
  Interventions: Drug: Somatropin
- Dehydroepiandrosterone (Experimental): DHEA 50 mg twice per day for 12 weeks in the last group , NATROL UK.Ltd.
  Interventions: Drug: Dehydroepiandrosterone

INTERVENTIONS:
Drug: myo-inositol — myo-inositol 600µgm + folic acid 0.2 mg) 2 capsules at the morning and 2 capsules at the evening on empty stomach for 12 weeks produced by a Lo.Li pharma international ,Rome.Italy .
  Other Names: Inofolic
  Arms: myo-inositol
Drug: Somatropin — growth hormone 2:Somatropin (4 IU for 1month), SEDICO ,6th of october .Egypt. 1 s.c injection every 3 days for at least 1 month.
  Arms: Somatropin
Drug: Dehydroepiandrosterone — DHEA 50 mg twice per day for 12 weeks in the last group , NATROL UK.Ltd.
  Other Names: DHEA
  Arms: Dehydroepiandrosterone

SUMMARY:
To evaulate the role of Myo-inositol, somatropin, DHEA on ICSI outcome in poor ovarian responder

DETAILED DESCRIPTION:
Each patient will be subjected to:

Full history taking. Systematic clinical examination to assess the general condition, body mass index (BMI) and local pelvic physical findings and AFC by trans-vaginal ultrasound on D2 to 3 of menstruation.

Routine labs as CBC, liver & kidney functions to exclude general disease as a contraindication for induction or pregnancy.

Blood sample will be obtained for assessment of basal serum levels of FSH, LH, E2 on days 2- 3 of the cycle. PRL, AMH and TSH Ovarian Stimulation The patients will begin injections of recombinant FSH (rFSH, Gonal-F; Merck-Serono, Italy) from day 2-3 of menstruation, with daily dose of 150-300 IU adjusted according to individual conditions on the basis of the antral follicle count (AFC),hormonal profile, age, body mass index (BMI), and previous ovarian response, according to the standard operating procedures of the center. .

For pituitary suppression, the patients will receive GnRH antagonist Cetrorelix (CETROTIDE 0.25Mg/d, Merck Serono, Germany) 0.25 mg/day subcutaneously from day 6 of induction until trigger day.

The serum LH, estradiol levels as well as number and size of follicles will be monitored every two days, starting from stimulation day 6 until the day of hCG injection.

ELIGIBILITY:
Inclusion Criteria:

* 1-Infertile women who have one of the criteria of poor ovarian response as follows ;
* Antral follicle count less than 7
* Anti-Mullerian hormone level Less than 1.2 ng/ml 2- females with body mass index (BMI) from 19-25

Exclusion Criteria:

1. Any endocrine or metabolic disorder such as polycystic ovary syndrome,
2. Hyperprolactinemia, diabetes and thyroid dysfunction.
3. Any pelvic pathology such as hydrosalpinx, uterine anomaly.
4. any male factor infertility such as Oligo-Astheno-Teratozoospermia (OAT) or Azoospermia.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Number and maturity of oocytes retrieved | 1 month
  Number and maturity of oocytes retrieved (M1/M2)

SECONDARY OUTCOMES:
chemical pregnancy rate | 1 month
  hcg positive

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No